CLINICAL TRIAL: NCT01555346
Title: A Clinical Study to Evaluate the Clinical Performance of the SEQureDx Trisomy 21 Test in the Detection of the Relative Quantity of Chromosome 21 in Circulating Cell-Free DNA Extracted From a Maternal Blood Sample Obtained From Pregnant Women With One or More High Risk Indicators for Fetal Chromosome 21 Aneuploidy
Brief Title: Clinical Evaluation of the SEQureDx T21 Test In High Risk Pregnancies
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-T21-304
Record Dates: First submitted 2012-02-15; First posted 2012-03-15 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Down Syndrome; Fetal Aneuploidy
Keywords: Down syndrome; fetal aneuploidy; trisomy; noninvasive prenatal test
MeSH Terms: conditions — Down Syndrome; Trisomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood specimens will be collected and processed to plasma. DNA will be extracted from the plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk pregnant subjects undergoing an invasive procedure: Women with one or more high risk factors for fetal chromosome 21 aneuploidy scheduled to undergo an invasive procedure for fetal karyotype determination.
- High risk subjects electing not to undergo invasive procedure: Women with one or more high risk factors for fetal chromosome 21 aneuploidy who elect not to undergo an invasive procedure for fetal karyotype determination.

SUMMARY:
Whole blood samples will be collected from high-risk pregnant women to validate the clinical performance of the SEQureDx Trisomy 21 Test.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman 18 years of age or older at 10 - 22 weeks gestation inclusive
* Subject has one or more high risk indicator for fetal chromosome 21 aneuploidy
* Subject provides signed and dated informed consent
* Subject agrees to provide a whole blood sample

Exclusion Criteria:

* Fetal demise at the time of the blood draw
* Previous specimen donation under this protocol

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between 10 and 22 weeks of gestation inclusive who have one or more high risk indicators for fetal chromosome 21 aneuploidy.
Sampling Method: Non-Probability Sample
Enrollment: 3062 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical Assay Performance | Performance of the assay will be based upon a single blood sample collected during the only study visit from a high risk pregnancy prior to the subject undergoing an invasive procedure (amniocentesis or CVS) to confirm fetal karyotype.
  Each subject will provide a single blood sample prior to undergoing an amniocentesis/CVS that will be processed to plasma and stored frozen until the end of the study. Frozen plasma samples will then be analyzed using the SEQureDx Trisomy Test and the sensitivity and specificity of the assay will be determined by comparing the plasma test results to the fetal karyotyping results obtained via aminiocentesis or CVS. A subject's participation ends after the results of the fetal karyotype are obtained and recorded.

SECONDARY OUTCOMES:
Subject selection bias assessment | A single blood sample will be collected at a single clinic visit from high risk pregnancies that refuse to undergo an invasive procedure.
  All subjects that enter the study are at high risk for fetal aneuploidy. However, sensitivity and specificity of the assay will be based upon those subjects that have a confirmed fetal karyotype obtained by amniocentesis/CVS. Subject selection bias assessment will be done by comparing SEQureDx Trisomy T21 Test results between women who agree to undergo an invasive procedure to obtain fetal karyotype and women who elect not to undergo an invasive procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Juan-Sebastian Saldivar, MD, Study Director — Sequenom Laboratories
Locations (29):
- United States (27):
  - University of South Alabama, Mobile, Alabama
  - Visions Clinical Research Tuscon, Tucson, Arizona
  - Obstetrix Medical Group of California, Campbell, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - San Gabriel Valley Perinatal Medical Center, Monterey Park, California
  - Scripps Clinic Carmel Valley, San Diego, California
  - South Florida Perinatal, Miami, Florida
  - Southeast Perinatal Associates - Miramar, Miramar, Florida
  - Southeast Perinatal Associates - Weston, Sunrise, Florida
  - Hawaii Pacific Health, Honolulu, Hawaii
  - University of Iowa Health Care, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Healthcare, Louisville, Kentucky
  - Willis-Knighton Physician Network, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Lukes Hospital of Kansas City, Kansas City, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Saint Peter's Hospital, New Brunswick, New Jersey
  - Virtua Health, Sewell, New Jersey
  - Virtua Health, Voorhees Township, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - Complete Healthcare for Women, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Regional Obstetrical Consultants, Chatanooga, Tennessee
  - Obstetrix Medical Group of Washington, Inc., Seattle, Washington
- Canada (2):
  - North York General Hospital, Toronto, Ontario
  - Chuq/Chul, Québec, Quebec

REFERENCES:
- [Background] Palomaki GE, Deciu C, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma reliably identifies trisomy 18 and trisomy 13 as well as Down syndrome: an international collaborative study. Genet Med. 2012 Mar;14(3):296-305. doi: 10.1038/gim.2011.73. Epub 2012 Feb 2. PMID 22281937
- [Background] Palomaki GE, Kloza EM, Lambert-Messerlian GM, Haddow JE, Neveux LM, Ehrich M, van den Boom D, Bombard AT, Deciu C, Grody WW, Nelson SF, Canick JA. DNA sequencing of maternal plasma to detect Down syndrome: an international clinical validation study. Genet Med. 2011 Nov;13(11):913-20. doi: 10.1097/GIM.0b013e3182368a0e. PMID 22005709
- [Background] Ehrich M, Deciu C, Zwiefelhofer T, Tynan JA, Cagasan L, Tim R, Lu V, McCullough R, McCarthy E, Nygren AO, Dean J, Tang L, Hutchison D, Lu T, Wang H, Angkachatchai V, Oeth P, Cantor CR, Bombard A, van den Boom D. Noninvasive detection of fetal trisomy 21 by sequencing of DNA in maternal blood: a study in a clinical setting. Am J Obstet Gynecol. 2011 Mar;204(3):205.e1-11. doi: 10.1016/j.ajog.2010.12.060. Epub 2011 Feb 18. PMID 21310373